CLINICAL TRIAL: NCT00922246
Title: Prevention of Lower Limb Overuse Injuries by Using Custom Made Insoles: A Randomized Controlled Trial of 230 Patients
Brief Title: Insoles in Prevention of Lower Limb Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Defense Forces (Other Government)
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 55555
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Lower Limb Overuse Injuries
Keywords: overuse injuries; conscript; prevention
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): Conscript used their own ankle boots instead of custom made insoles.
- shoe insoles (Experimental): The custom made insoles (Thermo+Camel, cost for the military 20,50 euros) were fabricated from firm-density polyethylene and the hard plastic shell was a three-quarter length. The insole was strong enough to fill the arch area thus providing support to the mid foot. It also influences the position of the foot. The insoles were individually customized by heating the polyethylene in form of individual foot with standing and walking in them. The conscripts were advised to use these insoles in their ankle boot.
  Interventions: Device: custom-made insoles (Thermo+Camel, cost for the military 20,50 euros)

INTERVENTIONS:
Device: custom-made insoles (Thermo+Camel, cost for the military 20,50 euros) — The custom made insoles (Thermo+Camel, cost for the military 20,50 euros) were fabricated from firm-density polyethylene and the hard plastic shell was a three-quarter length.
  Arms: shoe insoles

SUMMARY:
To address whether custom made foot insoles could be used for primary prevention of lower limb overuse injuries, the investigators conducted a prospective, randomized controlled study comparing the use of insoles and standard shoes in healthy young adults exposed to increased physical activity.

ELIGIBILITY:
Inclusion criteria:

* healthy conscripts without any diagnosed deformities of lower limb by physician in premilitary physical examination

Exclusion criteria:

* major orthopaedic or medical conditions (e.g., diabetes, inflammatory arthritis, previous severe trauma (exclusion criteria for the military service)
* patients were excluded from our study if they already had insoles prescribed by a physician or a physiotherapist (eight patients)
* since only 2% of Finnish conscripts are females, they were excluded from the study

Ages: 18 Years to 29 Years | Sex: Male
Age Groups: Adult
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The main outcome measure in the present study was a lower limb overuse injury requiring a visit at the garrison physician and requiring suspension from the duty. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Military Medicine, Helsinki, Finland